CLINICAL TRIAL: NCT05692544
Title: Image Data Collection of Tanned Skin During Phototherapy Treatment Using a Multi-spectral Camera
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUM-ABU-SMRT-22-03
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-04

CONDITIONS: Pigment; Lesion; Lesion; Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Phototherapy treatment — only patients was proscribe to phototherapy treatment can participate in the study

SUMMARY:
This is a prospective, observational, single-center, image collection study. Any patient who arrived at the phototherapy clinic for the first time, regardless of this study, and is prescribed a total of 30 treatments can be included, regardless of skin or medical condition.

After consenting subjects at least 5 close-up images will be taken from the specified anatomical areas, at different angles, using the SMART camera. Additional reference images of skin that is not exposed to the phototherapy treatment will be taken with the SMART Camera. Global image of the skin using a regular high-resolution camera is optional. The images will be collected on baseline visit, at least every 3 phototherapy treatments (approximately once a week), and at the last phototherapy treatment visit. i.e., in total of at least 11 phototherapy treatment visits. Follow-up images will be taken at 1-week and 2 weeks following the last phototherapy treatment.

Images shall be taken from any anatomical area that does not consist of any marked lesions or skin conditions. All images will be non-identifying.

DETAILED DESCRIPTION:
The SMART camera is advanced proprietary multi-spectral system camera, developed for research purposes. The SMART camera system is based on commercially available components and consists of 3 modules:

1. Camera Handpiece- Spectral module with a monochromatic camera, optics, and an array of LEDs at 7 different wavelengths.
2. Control Unit - an electronic box that powers and controls the camera. It includes electronics and a miniature computer.
3. Touch screen monitor - With user interface to operate the system When taking a photo, a series of cross-polarized monochromatic images are taken, each at different illumination color (wavelength). In total, seven images are taken with blue (450nm), teal (490nm), lime (570nm), orange (590nm), red (660nm), IR-1 (730nm), IR-2 (860nm). The total acquisition time for the seven images is 0.1sec. The images are stored in a dedicated directory on a removable hard disk in the control unit in correlation to patient ID entered through the user interface on the laptop. The number of images that can be taken is unlimited.

The camera passed the following safety tests by certified lab:

1. Check-up Safety Testing - IEC-60601-1 tests for investigational device by external laboratories according to IEC 60601-1, IEC 60601-2-22, IEC 60825-1, and IEC 60601-1-2 standards
2. LED Hazard Evaluation UV, Visible & NIR Test, according to IEC62471 by an external certified laboratory

ELIGIBILITY:
Inclusion Criteria:

* Any patient, male or female 18 years or older.
* Patient is scheduled for 30 treatments or more of phototherapy
* Subject is capable and willing to sign an informed consent
* Subject is willing to comply with study schedule
* Subject has areas of skin that do not consist any marked lesions, hairs or skin conditions and can be captured in the study

Exclusion Criteria:

• Subjects incapable of providing an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 10 subjects should be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Image data | 4-months
  Images will be collected through the study